CLINICAL TRIAL: NCT03805542
Title: Instillation of Renal Pelvis With 0.5% Iodophors for Patients With Calculous Pyonephrosis for I-stage PCNL : a Multicentre, Prospective, Open, Randomized Clinical Trial
Brief Title: Treatment of Calculous Pyonephrosis With 0.5% Iodophors for I-stage PCNL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Tj-czq8366
Record Dates: First submitted 2019-01-09; First posted 2019-01-15 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-07

CONDITIONS: Urolithiasis
Keywords: calculous pyonephrosis; I-stage PCNL; iodophors
MeSH Terms: conditions — Urolithiasis | interventions — Iodophors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): I-stage nephrostomy（Double J stent placement under cystoscopy） and II-stage operation
- I-stage operation group (Experimental): Disinfection of pelvis with 0.5% iodophors
  Interventions: Combination Product: 0.5% Iodophors

INTERVENTIONS:
Combination Product: 0.5% Iodophors — Before lithotripsy, 0.5% iodophor 40 ml(depending on the degree of hydronephrosis) was used to perfuse the calculous side pelvis under low pressure for 5 minutes.
  Arms: I-stage operation group

SUMMARY:
Calculous Pyonephrosis is a special type of urinary tract calculi, which is also common in clinical practice. If pyonephrosis is not treated in time, it will have a serious impact on the kidney function. Most stone operations can be performed in one stage, but there is still some controversy about whether PCNL can be performed in first stage for calculous pyonephrosis. The traditional idea is that nephrostomy should be performed first to induce pyuria caused by influenza, and then stone removal should be done in the second stage. However, I-stage nephrostomy and drainage and II-stage lithotripsy can also lead to prolonged hospitalization, increased medical costs and increased family burden. Based on the current treatment status of pyonephrosis patients, previous animal experimental results and volunteers' blood iodine absorption status, we intend to design a clinical trial of Stage-I percutaneous nephrolithotomy(PCNL) after iodophor disinfection of renal collecting system.

Iodophor, also known as povidone iodine, is composed of iodine and polyol ether surfactants. Iodophor disinfectant is a disinfectant with iodine as its main ingredient. It has strong bactericidal power and broad antimicrobial spectrum. It can kill viruses, bacterial propagules, fungi, protozoa, etc. 0.5% iodophor disinfectant (containing effective iodine 5000mg/L) can form a very thin bactericidal film on the wound surface and release it slowly and persistently.

At present, clinical studies on calculous pyonephrosis at home and abroad are mostly single-center, small sample studies, and lack of randomized controlled clinical trials. In view of the current situation and animal experimental results, we intend to carry out a clinical trial of "iodophor treatment of pyonephrosis and one-stage operation" in order to benefit patients with calculous pyonephrosis.

DETAILED DESCRIPTION:
Calculous Pyonephrosis is a special type of urinary tract calculi, which is also common in clinical practice. If pyonephrosis is not treated in time, it will have a serious impact on the kidney function. It can lead to renal failure and atrophy in the late stage. It can also cause acute peritonitis due to pus penetrating the renal capsule and endanger life. Most stone operations can be performed in first stage, but there is still some controversy about whether PCNL can be performed in first stage for calculous pyonephrosis. The traditional idea is that nephrostomy should be performed first to induce pyuria caused by influenza, and then stone removal should be done in the second stage. However, I-stage nephrostomy and drainage and II-stage lithotripsy can also lead to prolonged hospitalization, increased medical costs and increased family burden. With the widespread use of the third and fourth generation lithotripsy machines, ultrasound lithotripsy and lithotripsy system can reduce the pressure in drainage system, which makes more and more urologists begin to try one-stage surgical treatment for calculous pyonephrosis in non-acute infection period. Based on the current treatment status of pyonephrosis patients, previous animal experimental results and volunteers' blood iodine absorption status, we intend to design a clinical trial of Stage-I lithotripsy (PCNL) after iodophor disinfection of renal collecting system.

Iodophor, also known as povidone iodine, is composed of iodine and polyol ether surfactants. Iodophor disinfectant is a disinfectant with iodine as its main ingredient. It has strong bactericidal power and broad antimicrobial spectrum. It can kill viruses, bacterial propagules, fungi, protozoa, etc. 0.5% iodophor disinfectant (containing effective iodine 5000mg/L) can form a very thin bactericidal film on the wound surface and release it slowly and persistently. The principle of sterilization is to denaturate and precipitate proteins in pathogenic organisms, leading to inactivation of bacteria and other microorganisms, so as to achieve the purpose of efficient disinfection and sterilization.

It was found that the pharmacological action of iodophor solution containing 500 mg/L of available iodine was to release iodine gradually, which had the characteristics of low toxicity, little stimulation and long duration of pharmacodynamics. At present, 0.5% iodophor is widely used in skin disinfection before surgery, its effectiveness and safety are confirmed; intravenous drip of antibiotics one hour before surgery and 0.5% iodophor irrigation during operation can significantly reduce the incidence of wound infection after acute appendicitis surgery. In gynecological surgery, 0.5% iodophor is often used to disinfect vaginal mucosa, and effective anti-infective effect is achieved.

It was found that routine iodophor irrigation of wounds for 2-3 minutes during operation could effectively reduce the infection rate after operation, disinfect the skin area of operation field, and the effect of iodophor solution could last until the end of routine operation due to the slow release of iodine ions. Some researchers have studied the toxicology of iodophor disinfectant and found that: (1) the LD50 （Lethal Does,50%）value of animals tested in acute oral toxicity test is more than 5000mg/kg.bw, which is actually non-toxic; (2) multiple skin irritation tests are non-irritating; (3) acute eye irritation tests are non-irritating; (4) rabbit vaginal mucosa irritation index is extremely mild irritation; (5) subacute toxicity tests suggest hematology and there was no statistical difference between the blood biochemical indexes and the control group. Of course, people allergic to iodine preparations are not allowed to use them. At present, there are many reports about the application of iodophor solution in the disinfection of human mucosal tissues. Domestic studies have reported that bladder irrigation with 20 ml 0.5% iodophor in Intensive Care Unit(ICU) can prevent and treat bacterial and fungal infections in urinary tract. Foreign studies have shown that 0.2% povidone iodine can replace 1% silver nitrate for pelvic perfusion in chyluria patients (recurrence rate 9/22, or 22%; average follow-up 23.3 months). It should be noted that vaginal mucosal epithelium is a type of stratified flat epithelium, which belongs to human stratified epithelium. Its surface layer is flat cells with thick epithelium and has mechanical protective effect. The mucosal epithelium of renal pelvis, ureter, bladder and urethra is a kind of transitional epithelium (also known as metastatic epithelium), and also belongs to a kind of stratified epithelium. Its surface layer is columnar cells, because of the shape of these epithelial cells. The shape and hierarchy can change with the contraction or expansion of the organ, so they are named. Transitional epithelium is characterized by dense cytoplasm near the lumen and strong eosinophilic, forming a dark-stained shell, which can prevent the erosion of urine. Therefore, there are some similarities and differences between the two types of epithelium, which is of great significance for us to further study the application of iodophor in transitional epithelium. At present, clinical studies on calculous pyonephrosis at home and abroad are mostly single-center, small sample studies, and lack of randomized controlled clinical trials. In view of the current situation and animal experimental results, we intend to carry out a clinical trial of "iodophor treatment of pyonephrosis and I-stage operation" in order to benefit patients with calculous pyonephrosis.

ELIGIBILITY:
Inclusion Criteria:

1. Age (>18) at the time of admission;
2. Glomerular filtration rate (GFR) > 30 ml/min
3. Upper urinary tract calculi with ipsilateral pyogenic infection of renal collecting system
4. No fear of cold and fever or low temperature(<36°C) before operation;
5. According to the medical principle, PCNL treatment indications were given.
6. Leukocyte count was (4-12) 10^9/l. (Note: The above conditions should be met at the same time.)

Exclusion Criteria:

1. Complicated with severe cardiopulmonary and cerebrovascular diseases, coagulation dysfunction, hypertension, diabetes, etc.
2. iodine allergy;
3. lonely kidney or transplanted kidney;
4. Pregnancy patients;
5. those with hyperthyroidism, hypothyroidism or abnormal thyroid function;
6. Other matters that are taboo for operation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Estimated)
Dates: Start 2019-08 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of SIRS（Systemic inflammatory response syndrome） | Day 3
  Is there a statistical difference in the incidence of systemic inflammatory response syndrome between the control group and the experimental group?
Incidence of Urosepsis | Day 3
  Is there a statistical difference in the incidence of urosepsis between the control group and the experimental group?

CONTACTS AND LOCATIONS:
Overall Officials: Xinguang Wang, M.A., Principal Investigator — Ph.D. Postgraduates
Locations (1):
- Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No